CLINICAL TRIAL: NCT02246894
Title: An Open Multicentre Phase III Study to Investigate the Safety and Efficacy of Optivate® in Children Under 6 Years of Age With Severe Haemophilia A.
Brief Title: A Study to Investigate the Safety and Efficacy of Optivate® in Children Under 6 Years of Age With Haemophilia A.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bio Products Laboratory (Other)
Responsible Party: Sponsor
Other Study IDs: 8VWF05
Record Dates: First submitted 2014-09-02; First posted 2014-09-23 (Estimated); Last update posted 2018-02-15 (Actual); Status verified 2018-02

CONDITIONS: Haemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — optivate; Factor VIII

ARMS (1):
- Optivate® (Experimental): Optivate® (Human Coagulation Factor VIII)
  Interventions: Biological: Optivate® (Human Coagulation Factor VIII)

INTERVENTIONS:
Biological: Optivate® (Human Coagulation Factor VIII)

SUMMARY:
The main objectives of this study are:

* to assess Optivate® consumption (IU/kg consumed per month for prophylactic and on-demand therapy and dose at each bleed).
* to assess clinical outcome when treating a bleed with Optivate®.
* to evaluate Optivate® in terms of clinical tolerance and safety in children under the age of 6 years. .
* to assess FVIII inhibitor development during the study.

ELIGIBILITY:
Inclusion Criteria:

* Children under the age of 6 years with a diagnosis of severe Haemophilia A. Subjects who required FVIII therapy and did not demonstrate inhibitors to FVIII.

Children with history of inhibitors to FVIII or clinically significant renal or liver disease were not eligible to participate in the study.

Exclusion Criteria:

-

Max Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Start 2003-11; Primary Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
Consumption of FVIII | Day 0 to Week 26

CONTACTS AND LOCATIONS:
Locations (5):
- Poland (5):
  - Children's Haematology and Oncology Clinic, Ul., W. Chodzki Str., Lublin Voivodeship
  - Academic Children's Hospital, Children's Haematology and Oncology, Clinic 265 Wielicka str., Krakow
  - Specialist Centre for Medical Care of Mother and Children, Internal Ward 1, 7/8 Dr B. Krysiewicza str., Poznan
  - Department of Paediatrics, Haematology and Oncology, Medical University of Warsaw, 24 Marszalkowska str., Warsaw
  - Children's Clinic for Bone Marrow Transplant, Oncology and Haematology, Medical University of Wroclaw, 44 Bujwida str., Wroclaw

REFERENCES:
- See also: Related Info — http://www.bpl.co.uk